CLINICAL TRIAL: NCT04916015
Title: Comparative Study of the Histomolecular, Radiological and Prognostic Profiles Between Brain Gliomas of Children (0-14 Years) and Adolescents/Young Adults (15-25 Years) Treated in the Amiens University Hospital Between 2008 and 2020
Brief Title: Histomolecular Profiles of Gliomas in Children and Adolescent/Young Adults
Acronym: BioMol GLIOMA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2021_843_0062
Record Dates: First submitted 2021-06-01; First posted 2021-06-07 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Histological; Molecular Sequence Variation; Glioma
Keywords: Histological; Molecular; Glioma; adolescents/young adults; Children
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- children (0-14 years)
- AYAs (15-25 years)

SUMMARY:
In the last decades, many advances have been made in the field of genetic abnormalities of glial and glioneuronal brain tumors. In the 2016 World Health organization (WHO) Classification of Tumors of the Central Nervous System, the concept of "integrated" diagnosis emerged: histological and genetic/molecular features now define many entities. Since 2016, six updates have been published by the c-IMPACT-NOW (the Consortium to Inform Molecular and Practical Approaches to CNS Tumor Taxonomy- Not Official WHO) to develop and clarify the "integrated" diagnosis. In the future WHO 2021 Classification of Tumors of the Central Nervous System, "integrated" diagnoses will take up even more importance. Even if they can have similar histological features, gliomas of children are very different from the "adult" gliomas in the molecular mechanism of oncogenesis. The histomolecular features of adolescents/young adults (AYAs) can have similarities with "pediatric-type" or "adult-type" gliomas, but few studies have focused specifically on the histomolecular profiles of gliomas in AYAs.

The investigators would like to study the cohort of patients treated for a glial and glioneuronal tumor diagnosed under the age of 25 in the Amiens University Hospital between 2008 and 2020. The investigators would like to compare the histomolecular profiles of gliomas in children (0-14 years) and AYAs (15-25 years).

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient
* Patient treated in the Amiens University Hospital
* Patient treated for a glial or glioneuronal brain tumor according to the 2016 WHO Classification of Tumors of the Central Nervous System ("diffuse oligodendroglia or astrocytoma tumour," "another astrocytic tumor," "another glioma" or a "mixed neuronal or glioneuronal tumour").
* Diagnosis histologically confirmed or formally established by radiologist.
* Diagnosis established between January 1, 2008 and December 31, 2020.
* No patient opposition (from adult patient, or from the holder of parental authority of the minor patient).

Exclusion Criteria:

* Uncertain diagnosis
* Patient opposition (from adult patient, or from the holder of parental authority of the minor patient).

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: patients treated for a glial and glioneuronal tumor diagnosed under the age of 25 in the Amiens University Hospital between 2008 and 2020.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Histogical glioma differences between child group(0-14 years) and AYA group (15-25 years) | one year
Molecular glioma differences between child group(0-14 years) and AYA group (15-25 years) | one year

SECONDARY OUTCOMES:
Variation of glioma MRI profile between child group(0-14 years) and AYA group (15-25 years) | one year
  MRI profiles are EPI T2* MRI profiles

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No